CLINICAL TRIAL: NCT00138983
Title: Prevention of Glucocorticoid-Induced Osteoporosis in Patients With Rheumatic Diseases. The STOP-Study: a Randomized Placebo Controlled Trial With Alendronate Versus Alfacalcidol.
Brief Title: Prevention of Glucocorticoid-Induced Osteoporosis in Rheumatic Diseases: Alendronate Versus Alfacalcidol.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Health Care Insurance Board (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OG67-STOP-study
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2000-03

CONDITIONS: Rheumatoid Arthritis; Polymyalgia Rheumatica; Giant Cell Arteritis; Polymyositis; Wegener's Granulomatosis
Keywords: glucocorticoid-induced osteoporosis; rheumatic diseases; prevention; randomized double-blind, double placebo controlled trial; alendronate versus alfacalcidol
MeSH Terms: conditions — Arthritis, Rheumatoid; Polymyalgia Rheumatica; Giant Cell Arteritis; Polymyositis; Granulomatosis with Polyangiitis; Rheumatic Diseases

INTERVENTIONS:
Drug: Alendronate versus alfacalcidol (1-alpha OH vitamin D)

SUMMARY:
The purpose of this study is to determine wich treatment is the most effective in prevention of glucocorticoid-induced osteoporosis in patients with rheumatic diseases. The STOP-study: a randomized placebo controlled trial with alendronate versus alfacalcidol.

DETAILED DESCRIPTION:
Treatment with glucocorticoids (GCs) is associated with bone loss initiated already early in therapy, causing increased (vertebral) fracture risk. Bone loss is caused by inhibition of bone formation by GCs. Active vitamin D analogues like alfacalcidol directly stimulate osteoblasts leading to an increase in bone formation. Bisphosphonates like alendronate induce apoptosis of osteoclasts leading to inhibition of bone resorption.

We performed a randomized, double-placebo, double-blind clinical trial of 18 months duration in patients with a rheumatic disease, starting GCs in a dosage of 7.5 mg prednisone equivalent daily or higher. Two hundred one patients were allocated to receive either alendronate 10 mg and alfacalcidol-placebo daily or alfacalcidol 1 microgram and alendronate-placebo daily. Primary outcome was change in bone mineral density of the lumbar spine in 18 months, secondary outcome incidence of (symptomatic) morphometric vertebral deformities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a rheumatic disease.
* Starting treatment with glucocorticoids in a dosage of 7.5 mg prednisone equivalent daily or higher.
* All ethnic groups and races.

Exclusion Criteria:

* Glucocorticoid treatment in the past 12 months (except for 12 weeks preceding the study)
* Primary hyperparathyroidism, hyperthyroidism or hypothyroidism in last year
* Metabolic bone disease
* Creatinine clearance of < 50 ml/min
* Documented hypercalcemia or hypercalciuria, nephrolithiasis in the last 5 years
* Pregnancy or lactation
* Treatment in the last 12 months with hormone-replacement therapy
* Anabolic steroids, calcitonin, active vitamin D3 analogues, fluoride or bisphosphonates.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2000-05; Study Completion 2003-11

PRIMARY OUTCOMES:
Percent change in bone mineral density of the lumbar spine (lumbar vertebrae 2 to 4) at 18 months.

SECONDARY OUTCOMES:
Percent change in bone mineral density of the femoral neck and total hip at 18 months and incidence of morphometrical vertebral deformities, symptomatic vertebral fractures and non-vertebral fractures.

CONTACTS AND LOCATIONS:
Overall Officials: J.W.J. Bijslma, Prof., Principal Investigator — UMC Utrecht; R.N.J.T.L. de Nijs, MD, Study Director — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Lukert BP, Raisz LG. Glucocorticoid-induced osteoporosis: pathogenesis and management. Ann Intern Med. 1990 Mar 1;112(5):352-64. doi: 10.7326/0003-4819-112-5-352. PMID 2407167
- [Background] de Nijs RN, Jacobs JW, Algra A, Lems WF, Bijlsma JW. Prevention and treatment of glucocorticoid-induced osteoporosis with active vitamin D3 analogues: a review with meta-analysis of randomized controlled trials including organ transplantation studies. Osteoporos Int. 2004 Aug;15(8):589-602. doi: 10.1007/s00198-004-1614-5. Epub 2004 May 7. PMID 15138667
- [Background] Saag KG, Emkey R, Schnitzer TJ, Brown JP, Hawkins F, Goemaere S, Thamsborg G, Liberman UA, Delmas PD, Malice MP, Czachur M, Daifotis AG. Alendronate for the prevention and treatment of glucocorticoid-induced osteoporosis. Glucocorticoid-Induced Osteoporosis Intervention Study Group. N Engl J Med. 1998 Jul 30;339(5):292-9. doi: 10.1056/NEJM199807303390502. PMID 9682041
- [Result] de Nijs RN, Jacobs JW, Lems WF, Laan RF, Algra A, Huisman AM, Buskens E, de Laet CE, Oostveen AC, Geusens PP, Bruyn GA, Dijkmans BA, Bijlsma JW; STOP Investigators. Alendronate or alfacalcidol in glucocorticoid-induced osteoporosis. N Engl J Med. 2006 Aug 17;355(7):675-84. doi: 10.1056/NEJMoa053569. PMID 16914703
- [Derived] de Nijs RN, Jacobs JW, Lems WF, Laan RF, Algra A, Huisman AM, Buskens E, de Laet CE, Oostveen JC, Geusens PP, Bruyn GA, Dijkmans BA, Bijlsmat JW. [Alendronate more effective than alfacalcidol in the prevention of osteoporosis in patients with rheumatic disease who are starting glucocorticoid therapy]. Ned Tijdschr Geneeskd. 2007 May 26;151(21):1178-85. Dutch. PMID 17557758
- [Derived] Jacobs JW, de Nijs RN, Lems WF, Geusens PP, Laan RF, Huisman AM, Algra A, Buskens E, Hofbauer LC, Oostveen AC, Bruyn GA, Dijkmans BA, Bijlsma JW. Prevention of glucocorticoid induced osteoporosis with alendronate or alfacalcidol: relations of change in bone mineral density, bone markers, and calcium homeostasis. J Rheumatol. 2007 May;34(5):1051-7. Epub 2007 Apr 1. PMID 17407214